CLINICAL TRIAL: NCT01919827
Title: Treatment of Idiopathic Pulmonary Fibrosis With Bone Marrow Derived Mesenchymal Stem Cells
Brief Title: Study of Autologous Mesenchymal Stem Cells to Treat Idiopathic Pulmonary Fibrosis
Acronym: CMM/FPI
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CMM/FPI
Record Dates: First submitted 2013-08-01; First posted 2013-08-09 (Estimated); Last update posted 2018-05-03 (Actual); Status verified 2018-05

CONDITIONS: Idiopathic Pulmonary Fibrosis
Keywords: Idiopathic pulmonary fibrosis; Stem cells; Mesenchymal stem cells
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MSC endobronchial infusion (Experimental)
  Interventions: Biological: Endobronchial infusion of adult mesenchymal stem cells; Biological: Autologous mesenchymal stem cells derived from bone marrow

INTERVENTIONS:
Biological: Endobronchial infusion of adult mesenchymal stem cells
Biological: Autologous mesenchymal stem cells derived from bone marrow

SUMMARY:
Clinical Trial Phase I, open, multicentric, non randomized, study with escalating doses, to evaluate the safety and feasibility of treatment with mesenchymal stem cells in patients with diagnosis of idiopathic pulmonary fibrosis.

Primary endpoint: The aim is to evaluate the safety and feasibility of the endobronchial administration of mesenchymal autolog stem cells derived from bone marrow (BM-MSC)in patients with mild-to-moderate idiopathic pulmonary fibrosis.

Secondary endpoint:Assess the possible effect of the infusion of BM-MSC in stopping the fall of pulmonary function in patients with mild-to-moderate idiopathic pulmonary fibrosis.

ELIGIBILITY:
INCLUSION CRITERIA:

1. Capacity for signing informing consent and express the willing to fulfill all the requirements of the study protocol during the study.
2. The patients should be, in the researcher opinion, capable to fulfill all the requirements of the trial.
3. Male or female patients, 30 to 80 years old, inclusive.
4. Diagnosis of idiopathic pulmonary fibrosis according to the following criteria, based on the ATS/ERS Guidelines:

   1. Definite or probable usual interstitial pneumonia confirmed by surgical lung biopsy.
   2. In the absence of surgical lung biopsy, all the following:

   i. High resolution CT (HRCT) showing definite findings for idiopathic pulmonary fibrosis (FPI): bibasal reticular opacities with minimal ground glass opacities.

   ii. Absence of other known causes of FPI including toxicity from drugs, environmental exposure or connective tissue diseases.

   iii. Pulmonary function tests showing ventilatory restrictive pattern and/or impaired gas exchange (FVC and/or DLCO <90% of predicted)
5. FVC ≥ 50% of predicted value with ratio of FEV1 to FVC ≥ 0.70.
6. DLco (corrected for hemoglobin) ≥ 35% predicted value.
7. Capability of performing a 6 minutes walk test at the time of inclusion.

EXCLUSION CRITERIA:

Any of the following:

1. Current pregnancy or lactation.
2. Findings that are diagnostic of an interstitial pneumonia or restrictive respiratory disease condition other than UIP.
3. Obstructive pulmonary disease defined by FEV1/FVC < 0,7 or significant emphysema on HRCT.
4. Evidence of sustained improvement in FPI defined by improvement of respiratory function tests before inclusion, observed in >=2 test over the year prior to inclusion.
5. Active or recent respiratory infection (less than 60 days before inclusion) or history of frequent exacerbations of IPF from an infectious cause (more than 2/year over the last 2 years)
6. Hospitalization in the 60 days prior to inclusion due to acute exacerbation of IPF.
7. Chronic cardiac failure (functional class NYHA III/IV) or left ventricular ejection fraction < 25%.
8. Chronically receiving corticosteroid more than 10 mg of prednisone or equivalent, immunosuppressors or antifibrotic agents, including pirfenidone, D-penicillamine, colchicine, ciclosporin A, TNF-alpha antagonists, imatinib, IFN-gamma, azathioprine, cyclophosphamide, within the 30 days prior to inclusion.
9. The patient requires hemodialysis, peritoneal dialysis or hemofiltration.
10. History of malignancy, with the exception of skin squamous or basocellular carcinoma or cervix in situ carcinoma treated successfully.
11. History of ethanol abuse within the year prior to inclusion
12. The patient is participating in a clinical trial which includes other drugs or research products within the 28 days prior to baseline assessment.
13. Comorbidities limiting life expectancy to less than 12 months from the baseline assessment.
14. Medical or psychiatric condition serious or active which might interfere with the treatment of study, assessment or protocol fulfillment.
15. Positive test for HBsAg, HCV antibody, syphilis screening essays, or HIV antibody at screening.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2013-03; Primary Completion 2018-05-01 (Actual); Study Completion 2018-05-01 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse side effects. | Up to 12 months
  Number of participants with adverse side effects, and according to the level of severity:
  1. Low level: Increase in cough, fever or skin reactions
  2. Medium level: Infections not requiring hospital admission, mild alterations of renal or liver function
  3. High level: Death or major side effects requiring hospitalization:
     1. Worsening dyspnea with >=10% reduction in forced vital capacity, reduction in arterial pressure oxygen >= 10 mmHg and radiology progression between 3 months separated visits.
     2. Need for hospitalization due to respiratory failure requiring mechanical ventilation, worsening in gases exchange or lung infection.
     3. Carcinogenesis at 12 months after the endobronchial infusion of mesenchymal stem cells.

SECONDARY OUTCOMES:
Efficacy of the infusion of mesenchymal stem cells in stopping the fall in pulmonary function in patients with mild to moderate IPF | Up to 12 months
  Measures of efficacy:
  1. Fall in forced vital capacity as a continuous variable
  2. Progression of the disease defined by: Death, need for transplantation or deterioration in pulmonary function defined by fall in forced vital capacity (FVC) > 10% or in lung diffusion capacity (DLCO) > 15%.

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Servicio de Neumología, Clínica Universidad de Navarra, Pamplona, Navarre
  - Servicio de Neumología. Hospital Universitario de Salamanaca, Salamanca

REFERENCES:
- [Derived] Campo A, Gonzalez-Ruiz JM, Andreu E, Alcaide AB, Ocon MM, De-Torres J, Pueyo J, Cordovilla R, Villaron E, Sanchez-Guijo F, Barrueco M, Nunez-Cordoba J, Prosper F, Zulueta JJ. Endobronchial autologous bone marrow-mesenchymal stromal cells in idiopathic pulmonary fibrosis: a phase I trial. ERJ Open Res. 2021 Jun 28;7(2):00773-2020. doi: 10.1183/23120541.00773-2020. eCollection 2021 Apr. PMID 34195252